CLINICAL TRIAL: NCT07331454
Title: Robot-Assisted Versus Laparoscopy-Assisted Gastrectomy in Patients With cT4a Gastric Cancer: A Multicenter, Randomized Controlled, Phase III Study
Brief Title: Robotic vs Laparoscopic Gastrectomy for cT4a Gastric Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Affiliated Jiangning Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rosetta
Record Dates: First submitted 2025-12-28; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer (GC)
Keywords: gastric cancer; robotic gastrectomy; laparoscopic gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, superiority, open-label, multicenter randomized controlled trial. After central eligibility confirmation, participants are allocated 1:1 to robot-assisted or laparoscopy-assisted radical gastrectomy via a web-based block-randomization system stratified by center and intended extent of gastrectomy (distal vs total). Both arms receive standardized D2 lymph-node dissection aiming for R0 resection; post-operative care and adjuvant chemotherapy are delivered per local guidelines and recorded prospectively. Surgeons must hold ≥ 40 independent robotic/laparoscopic gastrectomy credentials, and operative videos are reviewed quarterly to ensure protocol fidelity. Cross-over is not permitted; conversion to open surgery is captured as a secondary safety endpoint. The model allows direct comparison of long-term oncologic efficacy while preserving pragmatic surgical and oncologic practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Gastrectomy (Experimental): Participants undergo radical gastrectomy (distal or total) performed with the da Vinci robotic system, including standardized D2 lymph-node dissection, aiming for R0 resection. All operative steps (lymph-node dissection, vessel ligation, digestive reconstruction) are completed with robotic instrumentation under 3-D high-definition vision and tremor-filtered wristed instruments.
  Interventions: Procedure: Robotic Gastrectomy
- Laparoscopic Gastrectomy (Active Comparator): Participants undergo the identical radical gastrectomy procedure (distal or total) performed with conventional laparoscopic instruments, including the same mandatory D2 lymph-node dissection and R0 resection criteria.
  Interventions: Procedure: Laparoscopic Gastrectomy

INTERVENTIONS:
Procedure: Robotic Gastrectomy — Radical gastrectomy (distal or total) performed with the da Vinci robotic system, including standardized D2 lymph-node dissection, aiming for R0 resection. All operative steps (lymph-node dissection, vessel ligation, digestive reconstruction) are completed with robotic instrumentation under 3-D high-definition vision and tremor-filtered wristed instruments.
  Arms: Robotic Gastrectomy
Procedure: Laparoscopic Gastrectomy — Radical gastrectomy procedure (distal or total) performed with conventional laparoscopic instruments, including the same mandatory D2 lymph-node dissection and R0 resection criteria.
  Arms: Laparoscopic Gastrectomy

SUMMARY:
The goal of this multicenter, randomized, phase III clinical trial is to test whether robot-assisted radical gastrectomy improves 3-year recurrence-free survival versus laparoscopy-assisted radical gastrectomy in adults aged 18-80 years with previously untreated, resectable cT4a gastric adenocarcinoma and non-bulky lymph nodes; the main questions are whether the robotic approach confers superior RFS and maintains equivalent peri-operative safety (Clavien-Dindo ≥ II complications) and better secondary oncologic outcomes, and participants will be randomized 1:1 to undergo standardized D2 resection via robotic or laparoscopic technique and followed for 5 years with scheduled recurrence, survival, and quality-of-life assessments.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed gastric or Siewert type III (and selected type II) gastro-oesophageal junction adenocarcinoma, clinical stage cT4a without bulky lymph-node enlargement on contrast-enhanced CT or MRI No prior neoadjuvant chemotherapy, radiotherapy, or other anti-cancer therapy Tumour deemed amenable to R0 resection by a board-certified gastric surgeon and radiologist ECOG performance status 0-1 Estimated life expectancy ≥ 6 months

Adequate organ function defined by:

* ANC ≥ 1.2 × 10⁹/L, platelet ≥ 100 × 10⁹/L, Hb > 8 g/dL (no transfusion/G-CSF within 14 days)
* ALT/AST ≤ 2.5 × ULN, total bilirubin ≤ 1.5 × ULN (or isolated indirect hyperbilirubinaemia)
* Serum creatinine ≤ 1.5 × ULN and calculated creatinine clearance ≥ 60 mL/min
* INR or PT ≤ 1.5 × ULN (therapeutic low-dose anticoagulation allowed)
* TSH and free T4 within normal limits or clinically insignificant deviation BMI ≥ 18.5 kg/m² or body weight ≥ 40 kg Signed informed consent

Exclusion Criteria:

cT4b disease, distant metastasis, or peritoneal cytology positive for malignancy Bulky lymph-node conglomerates (> 3 cm short axis) or N3 disease precluding D2 dissection Previous gastrectomy or major upper-abdominal surgery (except uncomplicated laparoscopic cholecystectomy) within 5 years Concurrent malignancy within 5 years (except adequately treated basal-cell carcinoma, carcinoma in situ, or stage I tumours) Gastric cancer arising from emergency presentation (bleeding, perforation, obstruction) Planned multi-visceral resection for non-oncologic indication Active bleeding diathesis; INR > 1.5 off anticoagulants; history of grade ≥ 3 bleeding within 4 weeks Arterial or venous thrombo-embolic event within 6 months Clinically significant cardiovascular disease: NYHA class III-IV heart failure, LVEF < 50 %, myocardial infarction or unstable arrhythmia within 6 months, QTc ≥ 450 ms (men) or ≥ 470 ms (women) Severe chronic pulmonary disease: FEV₁ < 50 % predicted or oxygen-dependent Uncontrolled diabetes (HbA1c > 8 %), active autoimmune disease requiring systemic immunosuppression, or corticosteroids > 10 mg/day prednisone equivalent within 14 days Active infection requiring systemic antibiotics, HIV, hepatitis B (HBV DNA ≥ 500 copies/mL), hepatitis C, or tuberculosis Pregnancy, lactation, or fertile participants unwilling to use effective contraception Psychological disorder, substance abuse, or any condition that, in the investigator's opinion, would compromise protocol compliance or safety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
RFS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China